CLINICAL TRIAL: NCT05781230
Title: The Effect of Exercises of Different Intensity Applied After Total Knee Arthroplasty on Exercise-Induced Hypoalgesia: Randomised Controlled Trial
Brief Title: The Effect of Exercises of Different Intensity Applied After Total Knee Arthroplasty on Exercise-Induced Hypoalgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, MERVE KARAPINAR, Assistant Professor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 126
Record Dates: First submitted 2023-02-24; First posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Knee Osteoarthritis; Pain, Acute
Keywords: Total Knee Arthroplasty; Exercises intensity; pressure pain threshold; exercise-induced hypoalgesia
MeSH Terms: conditions — Osteoarthritis, Knee; Acute Pain

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients were block-randomized based on intensity of exercises. The randomization sequence was produced by an external investigator using a computer-generated randomization sequence (Microsoft Excel, Microsoft, Redmond, WA, USA) to generate either a 0 or 1, corresponding with high intensity exercises or low intensity exercises, respectively
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIE program (Experimental): HIE program ; High Intensity Exercises Program. 3 sets of 15 repetition
  Interventions: Behavioral: High Intensity Exercises Program; Behavioral: Low Intensity Exercises Program
- LIE Program (Experimental): Low Intensity Exercises program 2 sets of 8 repetition
  Interventions: Behavioral: High Intensity Exercises Program; Behavioral: Low Intensity Exercises Program

INTERVENTIONS:
Behavioral: High Intensity Exercises Program — HIE program consisted of ankle pump exercise, Quadriceps isometric exercise, Terminal extension exercise, Passive-active assistive-active range of motion exercise, Heel sliding exercise, Straight leg raise exercise. All exercises were performed for 3 sets of 15 repetitions.
Behavioral: Low Intensity Exercises Program — LIE program: LIE program was similar to the HIE program. Main differences from the HIE program was repetitions of exercises. All exercises were performed by the patients for 2 sets of 8 repetitions and CPM sessions lasted each exercises session. LIE program took thirty minutes while HIE program lasted sixty minutes. Exercise intensity was monitored using the rating of perceived exertion (RPE) scale, maintaining a range between 6 and 20 RPE (16). PRE< 8 indicates low intensity, PRE>14 indicates high intensity

SUMMARY:
The aim of this study was to investigate whether exercise-induced hypoalgesia (EIH) is present following exercise in patient after total knee arthroplasty (TKA) and if so, if it changes with exercise intensity. A repeated measures and single-blinded randomized study were done. Thirty-eight patients 24 hours after TKA were randomly assigned to either low intensity exercises (LIE) group or high intensity exercises (HIE) group. An exercise programs lasted for five days during the hospitalization period. Pain severity was assessed by Visual Analog Scale (VAS) (0-10 mm). Pressure pain thresholds (PPTs) were measured over quadriceps and biceps brachii and muscles immediately before and after exercise.

DETAILED DESCRIPTION:
Background: The aim of this study was to investigate whether exercise-induced hypoalgesia (EIH) is present following exercise in patient after total knee arthroplasty (TKA) and if so, if it changes with exercise intensity.

Methods : A repeated measures and single-blinded randomized study were done. Thirty-eight patients 24 hours after TKA were randomly assigned to either low intensity exercises (LIE) group or high intensity exercises (HIE) group. An exercise programs lasted for five days during the hospitalization period. Pain severity was assessed by Visual Analog Scale (VAS) (0-10 mm). Pressure pain thresholds (PPTs) were measured over quadriceps and biceps brachii and muscles immediately before and after exercise.

ELIGIBILITY:
Inclusion Criteria:

* Patients had undergone primary unilateral total knee replacement surgery
* Patients hospitalized for at least seven days were enrolled in this study.

Exclusion Criteria:

* Medically stable patients who used glucocorticoids or strong analgesic drugs
* Patients had post-traumatic OA, rheumatoid arthritis (RA), psoriatic arthritis, cognitive, hearing and visual problems Patients were diagnosed chronic pain condition were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
change of pain severity | admission to hospital service to discharge from hospital service, an average 5 days
  . The pain severity evaluated using a visual analogue scale (VAS; scored from 0, no pain, to 100, the worst pain ever).
Change of Pressure pain theshold | admission to hospital service to discharge from hospital service, an average 5 days
  Pressure pain threshold (PPTs) were assessed using a handheld pressure algo-meter

CONTACTS AND LOCATIONS:
Overall Officials: MERVE KARAPINAR, PT, Principal Investigator — RESEARCH ASSİSSTANT
Locations (1):
- Merve Karapinar, Isparta, Turkey (Türkiye)